CLINICAL TRIAL: NCT00547144
Title: A Phase I/II Trial of Intratumoral Dendritic Cell Immunotherapy in Combination With Gemcitabine and Stereotactic Radiosurgery in Unresectable Pancreatic Cancer
Brief Title: Phase I/II Intratumoral DC Immunotherapy With Gemcitabine & XRT in Unresectable Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: George Albert Fisher (Other)
Responsible Party: Sponsor-Investigator, George Albert Fisher, Associate Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PANC0003; 95935 (Other: Stanford University alternate IRB Number); 1454 (Other: Stanford IRB); NCT00568932 (obsolete NCT alias)
Record Dates: First submitted 2007-10-18; First posted 2007-10-22 (Estimated); Last update posted 2012-11-08 (Estimated); Status verified 2012-08

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine (Experimental)
  Interventions: Drug: Gemcitabine; Procedure: Dendritic Cell Immunotherapy

INTERVENTIONS:
Drug: Gemcitabine — 1000 mg/m2 intravenoulsy once a week according to protocol schedule
  Other Names: Gemzar
Procedure: Dendritic Cell Immunotherapy — The cells will be administered by intratumoral injection on 2 different days(at least 21 days apart)
  Other Names: DC Therapy; Dendritic Cell Therapy

SUMMARY:
To determine the safety, feasibility and appropriate dendritic cell dose to vaccinate patients with pancreas cancer

ELIGIBILITY:
Inclusion Criteria:1. Patients must have histologically or cytologically confirmed adenocarcinoma of the pancreas. The site of the primary lesion should be confirmed endoscopically, radiologically, or surgically to be in the pancreas.

2. Patients must be deemed unresectable due to involvement of critical vasculature, adjacent organ invasion, presence of metastasis, or other medical condition making surgical resection unfavorable.

3. Patients must have a primary or metastatic lesion measurable in at least one dimension by RECIST criteria within 4 weeks prior to entry of study 4. More than 4 weeks must have elapsed from the time of major surgery or completion of the last dose of chemotherapy, radiation therapy, investigational therapy and patients must adequately recover from these effects.

5. Life expectancy of >3 months. 6. Karnofsky performance status >70%. 7. Patients must have normal organ and marrow functions as defined below: absolute neutrophil count >1,500/mm3 platelets >70,000/mm3 total bilirubin <1.5 mg/dL AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal creatinine within normal institutional limits OR creatinine clearance >60mL/min/1.73 m2 for patients with creatinine levels above institutional normal.

albumin > 2.8 mg/dL 8. Patients must have adequate clotting function (platelet > 70k; INR<1.4; PTT<60).

9. Age >18 years. 10. The effects of DCs on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

11. No history of autoimmune diseases. 12. Ability to understand the study protocol and a willingness to sign a written informed consent document. Exclusion Criteria:1. Patients receiving anticoagulation therapy.

2. Patients who have received prior gemcitabine or radiation therapy to the pancreatic bed 3. Patients receiving any other investigational agents. 4. Patients with known brain metastases will be excluded because of their poor prognosis and because they often develop progressive neurological dysfunction that would confound the evaluation of neurological and other adverse effects.

5. Uncontrolled concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements.

6. Patients who test positive for Hepatitis B virus, Hepatitis C virus or HIV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2005-10; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
o evaluate the immune response of patients treated with this regimen based on the presence and characterization of tumor-infiltrating white blood cells.
Phase II: To determine the overall response rate for this regimen as determined by radiographic criteria.
Phase I: To establish the maximally tolerated dose (MTD) and dose limiting toxicities (DLT) of intratumoral autologous dendritic cell vaccination in combination with gemcitabine and stereotactic radiosurgery
To determine the time to tumor progression for this regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Edgar G Engleman, Principal Investigator — Stanford University; George Albert Fisher M.D. Ph.D., Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States